CLINICAL TRIAL: NCT00475917
Title: A Phase 1 Dose-Escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of XL844 Administered as a Single Agent and in Combination With Gemcitabine in Subjects With Advanced Malignancies
Brief Title: A Study of XL844 Administered as a Single Agent and in Combination With Gemcitabine in Adults With Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL844-002
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Cancer; Lymphoma
Keywords: Advanced malignancies; Solid tumor
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — Gemcitabine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: XL844; Drug: Gemcitabine

INTERVENTIONS:
Drug: XL844 — Gelatin capsules supplied as 5-mg, 25-mg, and 100-mg strengths; twice-weekly dosing.
Drug: Gemcitabine — once-weekly 30-minute IV infusion

SUMMARY:
The purpose of this study is to determine a safe dose of XL844 in combination with gemcitabine, how often it should be taken, and how well people with cancer tolerate the combination of gemcitabine and XL844.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a histologically confirmed advanced malignancy (solid tumor or lymphoma) that is metastatic or unresectable, and for which standard curative or palliative measures do not exist or are no longer effective, and there are no therapies known to prolong survival.
2. The subject has disease that is assessable by tumor marker, physical, or radiologic means.
3. The subject is ≥18 years old.
4. The subject has an ECOG (Eastern Cooperative Oncology Group) performance status of ≤2.
5. The subject has adequate organ and marrow function.
6. The subject has the capability of understanding the informed consent document and has signed the informed consent document.
7. Sexually active subjects (male and female) must use medically acceptable methods of contraception during the course of the study.
8. Female subjects of childbearing potential must have a negative pregnancy test at screening.
9. If a subject has received more than three prior regimens of cytotoxic chemotherapy, more than two biologic regimens, or more than 3000 cGy to >25% of his or her bone marrow, the investigator must discuss with the sponsor regarding subject suitability before enrollment.
10. The subject has had no other diagnosis of malignancy (unless non-melanoma skin cancer, in situ carcinoma of the cervix, or a malignancy diagnosed ≥5 years ago, and has had no evidence of disease for 5 years prior to screening for this study).

Exclusion Criteria:

1. The subject has received anticancer treatment (eg, chemotherapy, radiotherapy, immunotherapy, biologic therapy, investigational agent, or hormones) within 14 days prior to the first dose of study drug.
2. The subject has not recovered to Grade ≤1 from adverse events (AEs) due to investigational agents or other medications administered more than 30 days prior to the first dose of study drug.
3. The subject has received radiation to >25% of his or her bone marrow within 30 days of XL844 treatment.
4. The subject has a primary brain tumor or known brain metastases.
5. The subject has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. The subject is pregnant or breastfeeding.
7. The subject is known to be positive for the human immunodeficiency virus (HIV).
8. The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.
9. The subject has a known allergy or hypersensitivity to any of the components of the XL844 formulation or gemcitabine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of XL844 as a single agent and in combination with gemcitabine when administered orally to subjects with advanced malignancies | Assessed at each visit/periodic visits
Determine the Combination maximum tolerated dose and dose-limiting toxicities for XL844 alone and in combination with gemcitabine | Assessed at periodic visits
Evaluate plasma pharmacokinetics and estimate renal elimination of XL844 as a single agent and in combination with gemcitabine | Assessed at periodic visits

SECONDARY OUTCOMES:
(Exploratory:) Assess tumor response after repeated administration of XL844 in combination with gemcitabine in subjects with advanced malignancies | Assessed at periodic visits
Pharmacodynamic correlates of XL844 activity in tumor tissue | Assessed at periodic visits

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - M.D. Anderson Cancer Center, Houston, Texas